CLINICAL TRIAL: NCT01061450
Title: Effect of the Addition of Simvastatin to Enalapril in Hypertensive Individuals With Average Cholesterol Levels and Diastolic Dysfunction
Brief Title: Simvastatin and Diastolic Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brasilia Heart Study Group (Other)
Collaborators: Fundação de Amparo a Pesquisa do Distrito Federal (Unknown); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Andrei C Sposito, Heart Institute (InCor), University of São Paulo Medical School, São Paulo, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Statin_DD
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Diastolic Dysfunction; Hypertension
Keywords: Diastolic dysfunction; hypertension; Statins; ACE inhibitor; Echocardiography
MeSH Terms: conditions — Hypertension | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Simvastatin (Experimental): Simvastatin 80 mg/day
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — 80 mg once a day
  Other Names: Zocor
  Arms: Simvastatin
Drug: Placebo — 1 pill once a day
  Arms: Placebo

SUMMARY:
Diastolic dysfunction (DD) is an increasingly frequent condition in hypertensive individuals whose treatment remains unclear. Its presence is related to higher morbidity and mortality independent of blood pressure levels. The aim of this study is to investigate the additive effect of simvastatin on enalapril on DD in hypertensive patients with average cholesterol levels.

For this aim, hypertensive patients with DD and LDL-cholesterol <160 mg/dL will undergo a run-in phase to achieve a systolic blood pressure (SBP) <135 mmHg and diastolic blood pressure (DBP) <85 mmHg with enalapril. Hydrochlorothiazide could be added when need to achieve SBP or DBP control. Four weeks after reaching the optimum anti-hypertensive regimen patients will be randomized to receive 80 mg simvastatin or placebo for a period of 20 weeks. Echocardiograms will be performed before and after treatment with measurement of left atrial volume, conventional and tissue Doppler velocities in early diastole and late diastole. The evaluation of these will allow to identify changes of DD severity after treatment.

ELIGIBILITY:
Inclusion Criteria:

* men or postmenopausal women aged between 40 and 65 years old
* normal fasting blood glucose (<100 mg/dL) and glucose tolerance test (<140 mg/dL)
* waist circumference < 102 cm (men) or < 88cm (women)
* triglycerides <150 mg/dL, LDL cholesterol ≤ 160 mg/dl
* creatinine <1.2 mg/dL, sinus rhythm
* the presence of grade 1 or 2 of DD with an ejection fraction of left ventricle > 55%
* absence of myocardial ischemia during dobutamine stress echocardiography

Exclusion Criteria:

* thyroid dysfunction
* acute or chronic liver disease
* regular use of 3 or more antihypertensive drugs
* secondary hypertension
* symptoms or history of atherosclerotic disease
* valvular dysfunction
* LVH 14 and use of statins in the last 6 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-11; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Changes in E/A ratio and e' wave velocity | 20 weeks

SECONDARY OUTCOMES:
Changes in left atrium volume. | 20 weeks
Changes in left ventricular mass. | 20 weeks
Changes in e´/a´ waves ratio. | 20 weeks
Changes in mitral deceleration time. | 20 weeks
Changes in the ratio of mitral inflow velocity to annular relaxation velocity. | 20 weeks
Changes in mitral annulus systolic velocity | 20 weeks
Diastolic function reserve index measured at peak stress with dobutamine | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adenalva LS Beck, MD, Principal Investigator — InCor Heart Institute; Andrei C Sposito, MD, PhD, Study Chair — University of Brasilia Medical School, Brasilia, Brazil; Maria E Otto, MD, PhD, Principal Investigator — Instituto de Cardiologia do Distrito Federal, Brasilia, Brazil
Locations (1):
- Instituto de Cardiologia do Distrito Federal, Brasília, Federal District, Brazil

REFERENCES:
- [Derived] Beck AL, Otto ME, D'Avila LB, Netto FM, Armendaris MK, Sposito AC. Diastolic function parameters are improved by the addition of simvastatin to enalapril-based treatment in hypertensive individuals. Atherosclerosis. 2012 Jun;222(2):444-8. doi: 10.1016/j.atherosclerosis.2012.03.030. Epub 2012 Apr 3. PMID 22554359